CLINICAL TRIAL: NCT00605280
Title: A Phase 2/3 Randomized, Controlled, Double-Masked, Multi-Center, Comparative Trial, In Parallel Groups, To Compare The Safety And Efficacy Of Intravitreous Injections Of 0.3 Mg Pegaptanib Sodium (Macugen®), Given As Often As Every 6 Weeks For 2 Years, To Sham Injections In Subjects With Diabetic Macular Edema (DME) Involving The Center Of The Macula With An Open-Label Macugen Year 3 Extension.
Brief Title: A Multi-Center Trial To Evaluate The Safety And Efficacy Of Pegaptanib Sodium(Macugen) Injected Into The Eye Every 6 Weeks For Up To 2 Years For Macular Swelling Associated With Diabetes, With An Open-Label Macugen Year Extension.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A5751013; EOP1013H; NCT00148811 (obsolete NCT alias)
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2011-03-30 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Macular Edema Associated With Diabetes Mellitus
Keywords: randomized sham-controlled multicenter macular edema
MeSH Terms: interventions — Standard of Care; pegaptanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sham Control (Sham Comparator)
  Interventions: Drug: Standard of Care
- Macugen (Experimental)
  Interventions: Drug: Macugen

INTERVENTIONS:
Drug: Standard of Care — Clinicians decision to use optional laser therapy.
  Arms: Sham Control
Drug: Macugen — Intravitreal injection of Macugen 0.3mg/90ul every 6 weeks up to 2 years.
  Arms: Macugen

SUMMARY:
The purpose of the study is to test whether Macugen injected into the eye improves vision in more patients than the currently existing standard of care laser therapy. The safety of Macugen compared to standard of care laser will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* macular edema associated with diabetes
* visual acuity between 20/50 and 20/200

Exclusion Criteria:

* recent laser therapy in the eye
* recent signs of uncontrolled diabetes
* blood pressure worse than 160/100
* severe cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2005-09; Primary Completion 2009-11 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (69):
- United States (27):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, ‘Aiea, Hawaii
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Lynbrook, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, West Columbia, South Carolina
  - Pfizer Investigational Site, Abilene, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, McAllen, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Australia (2):
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, East Melbourne
- Austria (2):
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Vienna
- Brazil (3):
  - Pfizer Investigational Site, Gioania, Goiás
  - Pfizer Investigational Site, Porto Alegre
  - Pfizer Investigational Site, São Paulo
- Canada (2):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Montreal, Quebec
- Pfizer Investigational Site, Bogotá, Colombia
- Czechia (4):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Prague
- Pfizer Investigational Site, Glostrup Municipality, Denmark
- France (7):
  - Pfizer Investigational Site, Créteil, Cedex
  - Pfizer Investigational Site, Clermont
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Marsielle
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Paris
- Germany (6):
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Düsseldorf
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Tübingen
- Pfizer Investigational Site, Athens, Greece
- India (4):
  - Pfizer Investigational Site, Ahmedabad
  - Pfizer Investigational Site, Bangalore
  - Pfizer Investigational Site, Hyderabad
  - Pfizer Investigational Site, New Delhi
- Italy (3):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Udine
- Pfizer Investigational Site, Nijmegen, Netherlands
- Pfizer Investigational Site, Coimbra, Portugal
- Pfizer Investigational Site, Bloemfontein, South Africa
- Pfizer Investigational Site, Bern, Switzerland
- United Kingdom (2):
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Sheffield

REFERENCES:
- [Derived] Loftus JV, Sultan MB, Pleil AM; Macugen 1013 Study Group. Changes in vision- and health-related quality of life in patients with diabetic macular edema treated with pegaptanib sodium or sham. Invest Ophthalmol Vis Sci. 2011 Sep 29;52(10):7498-505. doi: 10.1167/iovs.11-7613. PMID 21896838
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Original protocol included 0.3, 0.03, and 0.003 milligram (mg) pegaptanib sodium and sham treatment groups; the 0.03 and 0.003 mg doses were removed, affected participants given option of receiving 0.3 mg injections of pegaptanib sodium or study withdraw. Later, participants who hadn't completed Year 2 were eligible to enroll in Year 3 extension.
Groups:
- 0.3 mg Pegaptanib Sodium: Intravitreal injection of pegaptanib sodium, 0.3 mg every 6 weeks up to 2 years. Eligible participants had option to enroll in Year 3, open-label, extension phase during which participants received intravitreal injections of pegaptanib sodium, 0.3 mg every 6 weeks for 1 year.
- 0.03 mg Pegaptanib Sodium: Intravitreal injection of pegaptanib sodium, 0.03 mg every 6 weeks was planned for up to 2 years. The 0.03 mg dose was removed and participants given option of receiving 0.3 mg injection of pegaptanib sodium every 6 weeks for 2 years or withdrawing from the study.
- 0.003 mg Pegaptanib Sodium: Intravitreal injection of pegaptanib sodium, 0.003 mg every 6 weeks was planned for up to 2 years. The 0.003 mg dose was removed and participants given option of receiving 0.3 mg injection of pegaptanib sodium every 6 weeks up to 2 years or withdrawing from the study.
- Sham: Standard of care and sham injection (the application of an empty barrel of a needleless syringe). Eligible participants had option to enroll in Year 3, open-label, extension phase during which participants received intravitreal injections of pegaptanib sodium, 0.3 mg every 6 weeks for 1 year.
Period: Year 1
Arm/Group | 0.3 mg Pegaptanib Sodium | 0.03 mg Pegaptanib Sodium | 0.003 mg Pegaptanib Sodium | Sham
Started | 145 | 22 | 7 | 143
Received 0.3 mg Treatment | 144 | 13 | 3 | 0
Completed | 126 | 11 | 6 | 124
Not Completed | 19 | 11 | 1 | 19
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Adverse Event | 3 | 1 | 1 | 5
Not completed — Physician Decision | 7 | 4 | 0 | 6
Not completed — Withdrawal by Subject | 2 | 4 | 0 | 4
Not completed — Other | 2 | 1 | 0 | 1
Not completed — Lost to Follow-up or Patient non-comply | 5 | 1 | 0 | 2
Period: Year 2
Arm/Group | 0.3 mg Pegaptanib Sodium | 0.03 mg Pegaptanib Sodium | 0.003 mg Pegaptanib Sodium | Sham
Started | 126 | 11 | 6 | 124
Received 0.3 mg Treatment | 126 | 3 | 2 | 0
Completed | 102 | 5 | 0 | 102
Not Completed | 24 | 6 | 6 | 22
Not completed — Adverse Event | 4 | 0 | 2 | 4
Not completed — Physician Decision | 11 | 6 | 4 | 11
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 4
Not completed — Other | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up or Patient non-comply | 4 | 0 | 0 | 2
Period: Year 3 Extension
Arm/Group | 0.3 mg Pegaptanib Sodium | 0.03 mg Pegaptanib Sodium | 0.003 mg Pegaptanib Sodium | Sham
Started | 46 | 0 | 0 | 54
Received 0.3 mg Treatment | 46 | 0 | 0 | 54
Completed | 38 | 0 | 0 | 45
Not Completed | 8 | 0 | 0 | 9
Not completed — Adverse Event | 2 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 5
Not completed — Other | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up or Patient non-comply | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 0.03 mg Pegaptanib Sodium: Intravitreal injection of pegaptanib sodium, 0.03 mg every 6 weeks was planned for up to 2 years. The 0.03 mg dose was removed and participants given option of receiving 0.3 mg injection of pegaptanib sodium every 6 weeks up to 2 years or withdrawing from study.
- 0.003 mg Pegaptanib Sodium: Intravitreal injection of pegaptanib sodium, 0.003 mg every 6 weeks was planned for up to 2 years. The 0.003 mg dose was removed and participants given option of receiving 0.3 mg injection of pegaptanib sodium every 6 weeks up to 2 years or withdrawing from study.
- Total: Total of all reporting groups
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham | 0.03 mg Pegaptanib Sodium | 0.003 mg Pegaptanib Sodium | Total
Number analyzed (Participants) | 145 | 143 | 22 | 7 | 317
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (9.2) | 62.4 (10.3) | 64.7 (8.6) | 57.3 (10.1) | 62.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 65 | 11 | 4 | 139
  Male | 86 | 78 | 11 | 3 | 178

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Greater Than or Equal to ≥10 Letter (or 2 Line) Improvement in Vision at 1 Year
Description: Refraction and best-corrected visual acuity (VA) measurements were performed using retro-illuminated, modified Ferris-Bailey Early Treatment Diabetic Retinopathy Study (ETDRS) charts
Time Frame: Baseline, Year 1
Population: Modified Intent-to-Treat (MITT)1 population:participants with at least 1 dose of study treatment who completed baseline VA, had at least 1 post baseline VA assessment within 1 year; 2 sites not analyzed due to Good Clinical Practice deviations; the 0.03 and 0.003mg pegaptanib arms not analyzed for efficacy. Last Observation Carried Forward (LOCF).
Measure: Number; unit: Participants
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 133 | 127
Participants | 49 | 25
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.0047, Cochran-Mantel-Haenszel — Adjusted for glycolated hemoglobin (HbA1c), systolic blood pressure (BP), diastolic BP, and baseline VA. Baseline values not carried forward for missing post-baseline data; Odds Ratio (OR) = 2.38, 95% CI 2-sided [1.32 to 4.30]

2. Secondary Outcome: Number of Participants With a ≥ 10 Letter (or 2 Line) Improvement in Vision at 2 Years
Description: Refraction and best-corrected VA measurements were performed using retro-illuminated, modified Ferris-Bailey ETDRS charts
Time Frame: Baseline, Year 2
Population: Full Analysis Set (FAS)2 population:participants who had same treatment for 102 weeks (pegaptanib sodium or sham on/before Week 96) with baseline VA assessment, who met the following: had at least 1 post baseline VA within 2 years, before entry into the Year 3 open-label extension phase, or before withdrawing from the study prior to Week 102. LOCF.
Measure: Number; unit: Participants
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 133 | 123
Participants | 51 | 37
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.1904, Cochran-Mantel-Haenszel; Adjusted for HbA1c, systolic BP, diastolic BP, and baseline VA. Baseline values were not carried forward for any missing post-baseline data; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.85 to 2.53]

3. Secondary Outcome: Number of Participants With a ≥ 15 Letter Improvement in Vision at 1 Year
Description: as for outcome 2
Time Frame: Baseline, Year 1
Population: MITT1 population. LOCF.
Measure: Number; unit: Participants
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 133 | 127
Participants | 22 | 13
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.2466, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.74 to 3.34]

4. Secondary Outcome: Number of Participants With a ≥ 15 Letter Improvement in Vision at 2 Years
Description: as for outcome 2
Time Frame: Baseline, Year 2
Population: FAS2 population. LOCF.
Measure: Number; unit: Participants
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 133 | 123
Participants | 30 | 18
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.1388, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.86 to 3.26]

5. Secondary Outcome: Number of Eyes With a 2 or More Step Increase in Degree of Retinopathy at 1 Year
Description: Retinopathy changes were monitored using fundus photography and fluorescein angiograph (FA) assessments. An Independent Reading Center, using trained graders, evaluated the presence of retinopathy using a modified 12-step version of the ETDRS Final Retinopathy Severity Scale, that ranged from step 1 (retinopathy level of 10 or 12) to step 12 (retinopathy level of 85A or 85B) where an increase in the step or retinopathy level indicated a worsening of the condition.
Time Frame: Baseline, Year 1
Population: Evaluable participants from MITT1 population. Only 1 eye per participant was assessed in this study. LOCF.
Measure: Number; unit: Eyes
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 98 | 97
Eyes | 4 | 12
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.0468, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.07 to 0.99]

6. Secondary Outcome: Number of Eyes With a 2 or More Step Decrease in Degree of Retinopathy at 1 Year
Description: Retinopathy changes were monitored using fundus photography and FA assessments. An Independent Reading Center, using trained graders, evaluated the presence of retinopathy using a modified 12-step version of the ETDRS Final Retinopathy Severity Scale, that ranged from step 1 (retinopathy level of 10 or 12) to step 12 (retinopathy level of 85A or 85B) where a decrease in the step or retinopathy level indicated an improvement.
Time Frame: Baseline, Year 1
Population: Evaluable participants from MITT1 population. Only 1 eye per participant was assessed in this study. LOCF.
Measure: Number; unit: Eyes
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 98 | 97
Eyes | 10 | 3
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.1124, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.90, 95% CI 2-sided [0.73 to 11.55]

7. Secondary Outcome: Number of Eyes With a 2 or More Step Increase in Degree of Retinopathy at 2 Years
Description: Retinopathy changes were monitored using fundus photography and FA assessments. An Independent Reading Center, using trained graders, evaluated the presence of retinopathy using a modified 12-step version of the ETDRS Final Retinopathy Severity Scale, that ranged from step 1 (retinopathy level of 10 or 12) to step 12 (retinopathy level of 85A or 85B) where an increase in the step or retinopathy level indicated a worsening of the condition.
Time Frame: Baseline, Year 2
Population: FAS2 population. Number of participants analyzed (N) = participants with evaluable data. Only 1 eye per participant was assessed in this study. LOCF.
Measure: Number; unit: Eyes
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 103 | 102
Eyes | 6 | 13
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.1788, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.16 to 1.42]

8. Secondary Outcome: Number of Eyes With a 2 or More Step Decrease in Degree of Retinopathy at 2 Years
Description: as for outcome 6
Time Frame: Baseline, Year 2
Population: as for outcome 7
Measure: Number; unit: Eyes
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 103 | 102
Eyes | 17 | 3
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.0048, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 5.12, 95% CI 2-sided [1.45 to 18.06]

9. Secondary Outcome: Change From Baseline in Mean VA Score at 1 Year
Description: Changes in VA monitored through refraction and best-corrected VA measurements using retro-illuminated, modified Ferris-Bailey ETDRS chart with participants at a 4-meter distance from chart. Distance VA expressed as an ETDRS score (number of letters correctly read) ranging from 0 to 60, where higher ETDRS scores represented better vision. Change from baseline for each patient equaled the visual acuity obtained at the observation minus the visual acuity at baseline.
Time Frame: Baseline, Year 1
Population: MITT1 population. LOCF.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 133 | 127
scores on a scale
  Baseline | 57.0 (8.85) | 57.5 (8.11)
  Change at 1 year | 5.2 (9.94) | 1.2 (11.77)
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.0040, ANCOVA; [statistical method as in outcome 2, analysis 1]; Least Squares (LS) Mean = 3.90, 95% CI 2-sided [1.25 to 6.54]

10. Secondary Outcome: Change From Baseline in Mean VA Score at 2 Years
Description: as for outcome 9
Time Frame: Baseline, Year 2
Population: FAS2 population. LOCF.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 133 | 123
Scores on a scale
  Baseline | 57.0 (8.85) | 57.4 (8.20)
  Change at Year 2 | 6.2 (10.58) | 1.7 (11.68)
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.0011, ANCOVA; Adjusted for HbA1c, systolic BP, diastolic BP, and baseline VA. Baseline values were not carried forward for any missing post baseline data; LS Mean = 4.57, 95% CI 2-sided [1.85 to 7.29]

11. Secondary Outcome: Number of Participants Requiring Focal or Grid Laser Treatment During Year 1
Description: Included focal laser coagulation, focal laser photocoagulation, panretinal laser photocoagulation, retinal laser coagulation, and retinal laser photocoagulation
Time Frame: 1 year
Population: MITT1 population
Measure: Number; unit: Participants
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 133 | 127
Participants | 31 | 53
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.0023, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.24 to 0.74]

12. Secondary Outcome: Number of Participants Requiring Focal or Grid Laser Treatment During Year 2
Description: as for outcome 11
Time Frame: 2 years
Population: FAS2 population
Measure: Number; unit: Participants
Arm/Group | 0.3 mg Pegaptanib Sodium | Sham
Number analyzed (Participants) | 133 | 123
Participants | 34 | 57
Statistical Analysis 1: Comparison: 0.3 mg Pegaptanib Sodium vs Sham; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.23 to 0.69]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Groups:
- 0.3 mg Pegaptanib Sodium: Intravitreal injection of pegaptanib sodium, 0.3 mg every 6 weeks from baseline up to 2 years. Includes participants randomized to 0.3 mg pegaptanib sodium and participants randomized to lower doses of pegaptanib sodium who then converted to 0.3 mg pegaptanib sodium; for participants who converted to 0.3 mg pegaptanib sodium, only events that occurred while receiving 0.3 mg pegaptanib sodium treatment are reported.
- 0.03 mg Pegaptanib Sodium: Intravitreal injection of pegaptanib sodium, 0.03 mg every 6 weeks was planned for up to 2 years. Events reported for participants after start of treatment, but before they converted to 0.3 mg pegaptanib sodium or withdrew from study.
- 0.003 mg Pegaptanib Sodium: Intravitreal injection of pegaptanib sodium, 0.003 mg every 6 weeks was planned for up to 2 years. Events reported for participants after start of treatment, but before they converted to 0.3 mg pegaptanib sodium or withdrew from study.
- Sham: Standard of care and sham injection (the application of an empty barrel of a needleless syringe) from baseline up to Year 2. Events reported for participants after start of sham, but before they converted to 0.3 mg pegaptanib sodium or withdrew from study.
- 0.3 mg Pegaptanib Sodium (Year 3): Participants who were originally randomized to pegaptanib sodium, 0.3 mg who enrolled in Year 3, open-label, extension phase during which participants received intravitreal injections of pegaptanib sodium, 0.3 mg every 6 weeks for 1 year.
- Sham Conversion (Year 3): Participants who were originally randomized to Sham who enrolled in Year 3, open-label, extension phase during which participants received intravitreal injections of pegaptanib sodium, 0.3 mg every 6 weeks for 1 year.
Arm/Group | 0.3 mg Pegaptanib Sodium | 0.03 mg Pegaptanib Sodium | 0.003 mg Pegaptanib Sodium | Sham | 0.3 mg Pegaptanib Sodium (Year 3) | Sham Conversion (Year 3)
Serious Adverse Events (participants affected / at risk) | 42/174 | 4/22 | 0/7 | 35/143 | 4/46 | 6/54
Other Adverse Events (participants affected / at risk) | 110/174 | 15/22 | 7/7 | 100/143 | 11/46 | 10/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3 mg Pegaptanib Sodium (N=174) | 0.03 mg Pegaptanib Sodium (N=22) | 0.003 mg Pegaptanib Sodium (N=7) | Sham (N=143) | 0.3 mg Pegaptanib Sodium (Year 3) (N=46) | Sham Conversion (Year 3) (N=54)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Caridiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 3 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diabetic retinal oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Intraocular pressure increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Iris neovascularisation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 0
Myocardial ishaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Ocular hypertension (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0
Overweight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 1
Polyp colorectal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Renal embolism (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 3 | 0 | 0 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3 mg Pegaptanib Sodium (N=174) | 0.03 mg Pegaptanib Sodium (N=22) | 0.003 mg Pegaptanib Sodium (N=7) | Sham (N=143) | 0.3 mg Pegaptanib Sodium (Year 3) (N=46) | Sham Conversion (Year 3) (N=54)
Anterior chamber flare (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 13 | 2 | 0 | 10 | 3 | 0
Conjunctival haemorrhage (Eye disorders) | 34 | 3 | 1 | 20 | 1 | 7
Conjunctivitis (Eye disorders) | 9 | 0 | 1 | 6 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 11 | 0 | 0 | 5 | 4 | 0
Diabetic retinal oedema (Eye disorders) | 18 | 0 | 0 | 24 | 0 | 0
Diabetic retinopathy (Eye disorders) | 10 | 0 | 2 | 16 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 20 | 5 | 2 | 11 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 20 | 3 | 0 | 13 | 0 | 0
Intraocular pressure increased (Investigations) | 29 | 2 | 2 | 9 | 3 | 3
Lacrimation increased (Eye disorders) | 9 | 0 | 0 | 4 | 0 | 0
Macular oedema (Eye disorders) | 16 | 2 | 1 | 17 | 3 | 4
Myodesopsia (Eye disorders) | 10 | 2 | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 13 | 0 | 0 | 11 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 20 | 2 | 0 | 10 | 0 | 0
Retinal aneurysm (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Retinal exudates (Eye disorders) | 11 | 0 | 0 | 8 | 0 | 0
Retinal haemorrhage (Eye disorders) | 10 | 0 | 0 | 15 | 0 | 0
Retinal neovascularisation (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 16 | 1 | 2 | 14 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 10 | 0 | 0 | 11 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.